CLINICAL TRIAL: NCT03675750
Title: Effects of Hyperprolactinemia Induced by Antipsychotic Drugs on Bone Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 201740089
Record Dates: First submitted 2018-06-08; First posted 2018-09-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: antipsychotic drugs; hyperprolactinemia; bone metabolism
MeSH Terms: conditions — Schizophrenia; Hyperprolactinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum bone alkaline phosphatase ,serum β-crosslaps and prolactin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed to assess the severities of hyperprolactinemia caused by antipsychotic drugs and the effects of the duration of hyperprolactinemia on bone metabolism in schizophrenia patients.

DETAILED DESCRIPTION:
Hyperprolactinemia is a common adverse effect of antipsychotic drugs. Studies have shown that hyperprolactinemia may affect bone metabolism through direct and indirect effects and increase the risk of osteoporosis and fracture.The investigators assess the duration, the severity of hyperprolactinemia and its effects on bone metabolism in schizophrenics taking antipsychotic drugs through analyzing the correlation between prolactin levels and biochemical markers of bone metabolism and the correlation between the duration of hyperprolactinemia and abnormal bone metabolism. Meanwhile, the investigators aims to obtain the boundary value of prolactin levels in patients with abnormal bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of the disease meets the ICD-10 diagnostic criteria for schizophrenia 2. Subjects Intend to use atypical antipsychotics 3. Age between 18 and 50 years of age

Exclusion Criteria:

* 1. Pregnant and breast feeding women 2. Abnormal lipid metabolism 3. The level of serum alanine aminotransferase or aspartate aminotransferase is two times higher than the upper limit of the normal 4. Patients with diabetes or impaired fasting glucose 5. The level of prolactin is higher than normal 6. Patients taking drugs that affect bone metabolism (e.g. selective serotonin reuptake inhibitors antidepressants, antiepileptic drugs) 7. The level of creatinine is 1.2 times higher than the upper limit of the normal value

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chinese outpatients or inpatients with schizophrenia
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Bone turnover biochemical markers | baseline ,4 weeks ,8 weeks，12 weeks and 26 weeks
  changes in the level of serum bone alkaline phosphatase ,serum β-crosslaps and from baseline to 4, 8, 12 and 26 weeks after enrollment

SECONDARY OUTCOMES:
serum prolactin | baseline ,4 weeks ,8 weeks，12 weeks and 26 weeks
  changes in the level of serum prolactin from baseline to 4, 8, 12 and 26 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: LiHua Wang, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China